CLINICAL TRIAL: NCT06048952
Title: Bariatrik Cerrahi Sonrası Müzik Terapinin Postoperatif Bulantı Kusmayı Azaltma ve Hasta Memnuniyeti Üzerine Etkisi
Brief Title: The Effect of Music Therapy After Bariatric Surgery on Postoperative Nausea Vomiting and Patient Satisfaction
Acronym: BSMusicPONV
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sibel Yilmaz Sahin (Other)
Responsible Party: Sponsor-Investigator, Sibel Yilmaz Sahin, Assistant Professor, Saglik Bilimleri Universitesi Gulhane Tip Fakultesi
Organization: Saglik Bilimleri Universitesi Gulhane Tip Fakultesi (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: BSMusicPONV
Record Dates: First submitted 2022-01-12; First posted 2023-09-21 (Actual); Last update posted 2023-12-15 (Actual); Status verified 2023-12

CONDITIONS: Bariatric Surgery
Keywords: bariatric surgery; music therapy; nausea and vomiting, postoperative; nursing care
MeSH Terms: conditions — Postoperative Nausea and Vomiting | interventions — Music Therapy

STUDY DESIGN:
Intervention Model Description: Intervention and Non Intervention Group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Music Therapy (Active Comparator): 30 Minutes before evaluate PONV at 2nd,4th,6th,12th,24th hours
  Interventions: Behavioral: Music Therapy
- No Intervention (No Intervention): No intervention performed PONV evaluated at 2nd,4th,6th,12th,24th hours

INTERVENTIONS:
Behavioral: Music Therapy — Huseyni maqam, Pentatonic music
  Arms: Music Therapy

SUMMARY:
In this study, it was planned to evaluate the effectiveness of the use of music therapy, which is a non-pharmacological method, in addition to pharmacological treatment in patients with PONV after bariatric surgery, whose application frequency is increasing in the treatment of obesity, and to determine its effect on patient satisfaction. The findings of this study are considered to be effective in preventing nausea and vomiting, providing patient comfort, increasing evidence-based nursing knowledge and increasing the quality of care.

DETAILED DESCRIPTION:
Postoperative nausea and vomiting (POBK) according to ASPAN (American Society of PeriAnesthesia Nurses) are Nausea and vomiting seen in the first 24 hours after surgery (1). While PONV is seen in 20-30% of patients after general anesthesia, this rate increases up to 80% in high-risk patients (2). PONV, which is the second most common postoperative complaint after pain, is a stressful and uncomfortable situation for patients, but it can cause serious complications. These complications are; dehydration, electrolyte imbalance, acid-base imbalance, pulmonary aspiration, pneumothorax, hypoxia, esophageal rupture, increased intracranial pressure, suture rupture, bleeding (3). Due to the long duration of general anesthesia and the use of high-dose opioids, the incidence of PONV is higher in some types of surgery (eg, abdominal surgeries) (4). Recent studies have shown that laparoscopic, gynecological and cholecystectomy surgeries are high-risk surgeries in terms of PONV (5).

While obesity ranks second among the preventable causes of death in the world, bariatric surgery is seen as the most effective method in the treatment of morbid obesity (6). Bariatric surgeries are surgeries that carry a high risk in terms of PONC, since they are abdominal surgery, performed under general anesthesia, and the laparoscopic method is preferred. Antiemetics can be used in high-risk patients after risk factors are determined to prevent PONV. However, due to complications, the effectiveness of the use of antiemetic drugs in the management of PONC remains limited (7). Published guidelines on PONC management recommend the use of non-pharmacological methods in addition to pharmacological treatment in patients at high risk for PONV. Some of the complementary methods used to prevent PONV are acupuncture, aromatherapy, acupressure, progressive relaxation exercises, hypnosis, massage, and music therapy (7). It has been reported in the literature that music therapy is a non-pharmacological nursing practice that is used to manage nausea-vomiting and the severity of symptoms, has no side effects, is easy to use (8). In addition, it has been noted that music therapy has positive effects on analgesic requirement, hospital stay, reducing fatigue and the use of antiemetic drugs (8). Çetinkaya's study to determine the effect of music on the severity of postoperative nausea and vomiting after laparoscopic cholecystectomy showed that listening to music reduces the severity of nausea and the frequency of nausea (9). According to a randomized controlled study conducted by Madson and Silverman in a group of 58 solid organ transplant patients, less nausea and vomiting were found in the music therapy group (10). In a study conducted by Nilsson et al. on hysterectomy patients who underwent general anesthesia in the intraoperative period, it was observed that music did not affect nausea and vomiting (11). In another study by Laurion and Fetzer, it was reported that music had no effect on PONV (12). In the fourth consensus guideline on the treatment of postoperative nausea and vomiting, it has been reported that music is not an effective prophylactic method for PONV, but this information is based on a single randomized controlled study (12,13). When the literature is examined, it has been determined that there is no common view on the use of music therapy as a complementary method in the management of PONV and more studies should be done on this subject.

ELIGIBILITY:
Inclusion Criteria:

* Cognitive functions are sufficient,
* Able to communicate in Turkish,
* Between the ages of 18-80,
* Patients who voluntarily participated in the study

Exclusion Criteria:

* Patients who did not volunteer for the study,
* Patients who underwent open surgery
* whose mother tongue is not Turkish

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2021-05-02 (Actual); Primary Completion 2021-10-14 (Actual); Study Completion 2021-10-14 (Actual)

PRIMARY OUTCOMES:
Postoperative Nausea and Vomiting | Postoperative 2nd hour
  Simplified postoperative nausea and vomiting impact scale consisting of two questions, there are four options for each question that can be scored 0, 1, 2, 3 points. The first question asks whether there is vomiting or retching, if so, the frequency, and the answers are "0" no, "1" once, "2" twice, "3" three or more times and have four choices. In the second question, it is questioned whether there is nausea (feeling of discomfort in the stomach and feeling like vomiting), whether the feeling of nausea, if any, affects your daily life activities such as getting out of bed, moving comfortably in bed, walking normally, or eating and drinking; The answers are "0" not much, "1" sometimes, "2" often or often, "3" always. The numerical value of the answers given to the first and second questions is added and the result is found. A score of five or more on the scale defines "clinically significant nausea and vomiting".
Postoperative Nausea and Vomiting | Postoperative 4th hour
  Simplified postoperative nausea and vomiting impact scale consisting of two questions, there are four options for each question that can be scored 0, 1, 2, or 3 points. The first question asks whether there is vomiting or retching, if so, the frequency and the answers are no, once, twice, three or more times and have four choices. In the second question, is questioned whether there is nausea (feeling of discomfort in the stomach and feeling like vomiting), whether the feeling of nausea, if any, affects your daily life activities such as getting out of bed, moving comfortably in bed, walking normally, or eating and drinking; The answers are not much, sometimes, often or often, always. The numerical value of the answers given to the first and second questions is added and the result is found. A score of five or more on the scale defines clinically significant nausea and vomiting.
Postoperative Nausea and Vomiting | Postoperative 6th hour
  Simplified postoperative nausea and vomiting impact scale consisting of two questions, there are four options for each question that can be scored 0, 1, 2, or 3 points. The first question asks whether there is vomiting or retching, if so, the frequency and the answers are no, once, twice, three or more times and have four choices. In the second question, is questioned whether there is nausea (feeling of discomfort in the stomach and feeling like vomiting), whether the feeling of nausea, if any, affects your daily life activities such as getting out of bed, moving comfortably in bed, walking normally, or eating and drinking; The answers are not much, sometimes, often or often, always. The numerical value of the answers given to the first and second questions is added and the result is found. A score of five or more on the scale defines clinically significant nausea and vomiting.
Postoperative Nausea and Vomiting | Postoperative 12th hour
  Simplified postoperative nausea and vomiting impact scale consisting of two questions, there are four options for each question that can be scored 0, 1, 2, or 3 points. The first question asks whether there is vomiting or retching, if so, the frequency and the answers are no, once, twice, three or more times and have four choices. In the second question, is questioned whether there is nausea (feeling of discomfort in the stomach and feeling like vomiting), whether the feeling of nausea, if any, affects your daily life activities such as getting out of bed, moving comfortably in bed, walking normally, or eating and drinking; The answers are not much, sometimes, often or often, always. The numerical value of the answers given to the first and second questions is added and the result is found. A score of five or more on the scale defines clinically significant nausea and vomiting.
Postoperative Nausea and Vomiting | Postoperative 24th hour
  Simplified postoperative nausea and vomiting impact scale consisting of two questions, there are four options for each question that can be scored 0, 1, 2, or 3 points. The first question asks whether there is vomiting or retching, if so, the frequency and the answers are no, once, twice, three or more times and have four choices. In the second question, is questioned whether there is nausea (feeling of discomfort in the stomach and feeling like vomiting), whether the feeling of nausea, if any, affects your daily life activities such as getting out of bed, moving comfortably in bed, walking normally, or eating and drinking; The answers are not much, sometimes, often or often, always. The numerical value of the answers given to the first and second questions is added and the result is found. A score of five or more on the scale defines clinically significant nausea and vomiting.

SECONDARY OUTCOMES:
Participant's satisfaction with the nursing care with | Postoperative 24th hour
  Numerical Rating scale consisting of numbers between "0" and "10" (0: not at all satisfied 10: very satisfied) have been used to determine the satisfaction level of patients at the 24th postoperative hour.

CONTACTS AND LOCATIONS:
Overall Officials: Sibel YILMAZ SAHIN, Asst.Prof., Principal Investigator — Saglik Bilimleri Universitesi Gulhane Tip Fakultesi
Locations (1):
- University of Health Sciences, Ankara, Turkey (Türkiye)